CLINICAL TRIAL: NCT06029088
Title: Risk-adapted Strategy Combining Magnetic Resonance Imaging and Prostate-specific Antigen Density to Individualize Biopsy Decision in Patients With PI-RADS 3 'Gray Zone' Lesions
Brief Title: Risk-adapted Strategy Including Magnetic Resonance Imaging and Prostate-specific Antigen Density in Blood for Biopsy Decision in Patients With Lesions Suspicious for Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Cagri Akpinar, M.D., Ankara Etlik City Hospital
Other Study IDs: I05-328-23
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate cancer; Risk-adapted strategy; Magnetic resonance imaging; Prostate-specific antigen density; PIRADS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent guidelines now recommend multi parametric magnetic resonance imaging prior to biopsy for all men as an integral part of improved diagnosis of clinical significant prostate cancer. However, magnetic resonance imaging targeted biopsy is a strategy that focuses on maximizing detection of clinical significant prostate cancer, but this procedure has the disadvantage of leading to higher detection of clinically insignificant prostate cancers. One of the risk-stratifications developed to minimize the existing disadvantages and avoid unnecessary biopsy procedures is a strategy in which multi parametric magnetic resonance imaging and prostate-specific antigen density are used in combination. This is especially important in all patients with PI-RADS (Prostate Imaging Reporting and Data System) 3 lesions which are also interpreted as indeterminate mpMRI findings. Current guidelines suggest that biopsy may be omitted in some patient groups with PI-RADS 3 lesions in the risk-adapted strategy involving prostate-specific antigen density. The aim of this study was to evaluate the role of risk-adapted strategies involving prostate-specific antigen density in biopsy decision to avoid unnecessary biopsy vs the risk of missing clinical significant prostate cancer diagnosis in patients with PI-RADS 3 lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who all had undergone multi parametric magnetic resonance imaging at our hospital
* Patients who all had undergone transrectal ultrasonography guided cognitive and fusion targeted biopsies

Exclusion Criteria:

* Magnetic resonance imaging at exterior hospitals
* Insufficient image quality/artifacts
* Previous prostate biopsy and/or prior prostate cancer diagnosis

Ages: 45 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Because prostate cancer is a male-specific disease
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Reducing unnecessary prostate biopsy with the combined use of magnetic resonance imaging and prostat-specific antigen density measurement | 2 weeks from the outpatient clinic admission

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)